CLINICAL TRIAL: NCT02346591
Title: Emotion Management Training: An Innovative Stress Reduction Program
Brief Title: Mobile-Web Emotion Self-management Tool
Acronym: Emotions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Principal Investigator, Amy Birney, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 102-2R
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Stress; Depression
Keywords: Positive psychology; Wellbeing; Stress reduction; Relaxation; Gratitude; Mobile app; Intervention; Altruism; Psychological well-being; Social well-being; Physical well-being; Workplace engagement
MeSH Terms: conditions — Depression; Altruism; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jauntly (Experimental): Mobile app designed to take advantage of the known connections between positive emotions, stress reduction and stress resilience; goal was to lead users through research-proven positive emotion enhancing exercises and relevant educational materials. Intervention activities covered five well-being generating content areas: 1) promoting the experience and recognition of gratitude; 2) encouraging positive social relationships and feelings of social support; 3) improving stress resilience via mindfulness and other relaxation-focused activities; 4) focusing and capitalizing on individual strengths (as opposed to limitations and weaknesses); and 5) general positive mood inducing activities.
  Interventions: Behavioral: Jauntly
- Online stress management information (Active Comparator): The control participants were emailed links to vetted online information about stress and encouraged to visit the websites.
  Interventions: Behavioral: Online stress management information

INTERVENTIONS:
Behavioral: Jauntly — Mobile app designed to encourage positive emotion-enhancing and stress reduction activities.
  Arms: Jauntly
Behavioral: Online stress management information — Online educational information about stress management
  Arms: Online stress management information

SUMMARY:
The investigators developed a responsive mobile-web app, "Jauntly," which was designed to take advantage of the known connections between positive emotions, stress reduction and stress resilience. The app's goal was to lead users through research-proven positive emotion-enhancing exercises and relevant educational materials. Intervention activities covered five well-being-generating content areas: 1) promoting the experience and recognition of gratitude; 2) encouraging positive social relationships and feelings of social support; 3) improving stress resilience via mindfulness and other relaxation-focused activities; 4) focusing and capitalizing on individual strengths (as opposed to limitations and weaknesses); and 5) general positive mood inducing activities. Program content was adapted from a variety of stress-relevant research areas including health psychology/psychosomatic medicine, social/personality psychology, positive psychology, and clinical psychology.

DETAILED DESCRIPTION:
The overarching goal of the Jauntly mobile app was to experience exercises that encourage one to take care of oneself emotionally, improve positive emotions, and decrease stress and other negative emotions. The user interacted with the app through evidence-based activities (e.g. writing gratefulness notes, helping others, practicing mindfulness). The activities were selected based on the goals the user selected upon initiation of program and throughout engagement with the app. In order to promote sustained use of the program and mastery of the positive emotion based skills, the design of the program included activities that range in difficulty so that the user could progress and improve (i.e., simple "1 and done" types of goals versus multi-week goals).

Research in positive psychology interventions suggests that increases in well-being are highest when the activity: 1) fits the person's interests and values and 2) is performed neither too frequently nor too seldom. Because of our desire to have a product with long-lasting usability and sustained engagement, it was critical that there were a diverse number of activities from which individuals could choose based on interest, current mood, and past success. The Jauntly user experience is structured around free use of the app partnered with regular emails, in-app messaging, videos, and articles. Emails remind users to utilize program content (including users in the control group who were reminded to visit the stress-management website). Use of the app and viewing of videos and other content is not restricted and users are able to self-tailor use according to their interest.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Employed at least part-time
* Self-report stress at work
* English speaking
* Access to a computer with high-speed internet connection, audio-video capability and an active email account

Exclusion Criteria:

* High level of self-reported grief
* High level of self-reported depression (PHQ-2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall perceived stress | 12 weeks
  The 10-item Perceived Stress Scale (PSS) assessed perceptions of feeling like you can not cope with things in your life and feelings of "stress" and nervousness on a scale of 1 (Never) to 5 (Very Often). The PSS is the most widely used self-report stress scale available, and has been shown to predict many important well-being outcomes.

SECONDARY OUTCOMES:
Psychological well-being assessed as positive and negative affect | 8 weeks, 12 weeks
  Positive and negative affect over the past few weeks was assessed at each time point using the Positive and Negative Affect Scale-expanded version, with a few nonrelevant items (e.g., surprise) removed, resulting in a total of 53 emotion adjectives on a scale of 1 (not at all/very slightly) to 5 (extremely). Subscales assessing positive affect (PA) and negative affect (NA) were created as well as specific basic emotion scales assessing fear (6 items), hostility (6 items), guilt (6 items), sadness (5 items), joviality (8 items), self-assuredness (6 items), attentiveness (4 items), fatigue (4 items) and serenity (3 items).
Self-reported depressive symptomatology | 8 weeks, 12 weeks
  Depressive symptomatology was assessed using the self-reported Center for Epidemiologic Studies Short Depression Scale (CESD-10). Participants are asked to rate each symptom on a scale of rarely/none of time to (1) to all of the time (4).
Self-reported social well-being | 8 weeks, 12 weeks
  The 10-statement UCLA Loneliness Scale asked users to respond to the root statement "How often do you feel…." in conjunction with various statements describing social relationships; e.g., "How often do you feel as if nobody really understands you?" Responses were on a 4-point scale (1-often; 4=never)
Self-reported physical well-being | 8 weeks, 12 weeks
  Eleven items were selected from the SF-36, a measure of functional status which contains 8 subscales. Items from 2 of the subscales were included: bodily pain and general health perceptions. Response scales were different for each of the subscales.
Workplace outcomes | 8 weeks, 12 weeks
  Absenteeism and presenteeism were assessed using the Workplace Outcomes Suite. A score from a 9-item work engagement assessment including questions about hours of missed work due to absenteeism, lateness, leaving early, and questions about lost productivity due to lack of concentration or personal distractions involving disrupting phone calls, email.
Users' perception of app usability | 8 weeks, 12 weeks
  Treatment participants completed the System Usability Scale, a quantitative measure of program ease of use (Sauro, 2011). The scale includes 10 items and users were asked to what degree they agreed or disagreed with program use and satisfaction statements on a 6-point scale (1=strongly disagree; 6=strongly agree).
User satisfaction with the app experience | 8 weeks, 12 weeks
  Users were asked 6 items pertaining to satisfaction and likelihood of continued use or recommendation of the Jauntly program specifically, on a 7-point scale (1=Not at all satisfied/likely; 7=Extremely satisfied/likely).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Birney, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States